CLINICAL TRIAL: NCT01970241
Title: Inpatient Diabetes on Corticosteroids
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hennepin Healthcare Research Institute (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MMRF-13-3658
Record Dates: First submitted 2013-09-04; First posted 2013-10-28 (Estimated); Results first posted 2019-10-01 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Diabetes Mellitus
Keywords: corticosteroid; diabetes; insulin
MeSH Terms: conditions — Diabetes Mellitus; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- NPH with steroid dose (Experimental): Receive NPH with each corticosteroid dose during the study duration (2-5 days).
  Low dose corticosteroids High dose corticosteroids Eating and 6a-8p 0.15 units NPH/kg 0.3 units NPH/kg NPO(nothing by mouth) or 8p-6a 0.1 units NPH/kg 0.2 units NPH/kg
  Interventions: Drug: NPH; Drug: Correction Factor
- Control - Background and correction insulin (Active Comparator): Receive usual care with background insulin and correction factor for duration of study (2-5 days)
  Interventions: Drug: Correction Factor

INTERVENTIONS:
Drug: NPH — NPH given per study table based on steroid dose and patient weight in kg.
  Other Names: NPH Lilly Insulin
  Arms: NPH with steroid dose
Drug: Correction Factor — Given at 2 units per 50 mg/dl over 200 mg/dl and increased to 3 units/50 mg/dl over 200 if glucose rises to over 300 mg/dl. Administered qid during study duration.
  Other Names: Rapid acting regular insulin

SUMMARY:
Despite a significant problem with out-of-control glucose levels in patients with diabetes receiving corticosteroids for a variety of illnesses, there are no published protocols addressing how to adequately treat corticosteroid-induced hyperglycemia. Investigators propose to test a protocol using scheduled dosing of NPH (Neutral protamine Hagedorn) insulin for inpatients with diabetes receiving corticosteroids. NPH insulin action is ideally timed to counteract corticosteroid-induced hyperglycemia, and the dose is added to the patient's usual insulin regimen and timed to correspond to the corticosteroid dosing regimen. Investigators will prospectively enroll eligible consented patients with diabetes who are receiving corticosteroids as part of their treatment in a large county hospital, will randomize them to intervention or control groups, and will monitor their glucose levels during their inpatient stay. The protocol will demonstrate improved control of glucose levels with minimal risk of hypoglycemia, and will provide a practical and readily implementable protocol using NPH insulin as therapy for corticosteroid-induced diabetes.

DETAILED DESCRIPTION:
As above.

ELIGIBILITY:
Inclusion Criteria:

* Prior history of diabetes
* Able to provide informed consent
* Receiving corticosteroids while hospitalized of greater than 10 mg/d prednisone or the equivalent of dexamethasone or methylprednisolone
* Expect to be hospitalized for 48 hours

Exclusion Criteria:

* Renal failure with GFR (glomerular filtration rate) < 30 ml/min/1.73m2
* ALT (alanine aminotransferase) > 2 times upper normal for laboratory

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2014-07; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Fish, MD, Principal Investigator — Hennepin County Medical Center, Minneapolis
Locations (1):
- Hennepin County Medical Center, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Khowaja A, Alkhaddo JB, Rana Z, Fish L. Glycemic Control in Hospitalized Patients with Diabetes Receiving Corticosteroids Using a Neutral Protamine Hagedorn Insulin Protocol: A Randomized Clinical Trial. Diabetes Ther. 2018 Aug;9(4):1647-1655. doi: 10.1007/s13300-018-0468-3. Epub 2018 Jun 30. PMID 29961246

RESULTS

PARTICIPANT FLOW:
Groups:
- NPH With Each Steroid Dose: Receive NPH with each corticosteroid dose during the study duration (2-5 days).
  Low dose corticosteroids eating: 0.2 units NPH/kg High dose corticosteroids eating: 0.3 units NPH/kg Low dose corticosteroids NPO: 0.1 units NPH/kg High dose corticosteroids NPO: 0.15 units NPH/kg
  NPH: NPH given per study table based on steroid dose and patient weight in kg.
  Correction Factor: Given at 2 units per 50 mg/dl over 200 mg/dl and increased to 3 units/50 mg/dl over 200 if glucose rises to over 300 mg/dl. Administered qid during study duration.
  Low dose corticosteroids: Prednisone 10 - 40 mg daily or equivalent corticosteroid dose.
  High dose corticosteroids: Prednisone > 40 mg daily or equivalent corticosteroid dose.
- Control: Receive usual care with background insulin and correction factor for duration of study (2-5 days)
  Correction Factor: Given at 2 units per 50 mg/dl over 200 mg/dl and increased to 3 units/50 mg/dl over 200 if glucose rises to over 300 mg/dl. Administered qid during study duration.
Period: Overall Study
Arm/Group | NPH With Each Steroid Dose | Control
Started | 46 | 39
Completed | 29 | 31
Not Completed | 17 | 8
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Steroid d/c;discharge<48 hrs. | 15 | 8

BASELINE CHARACTERISTICS:
Groups:
- NPH With Corticosteroid Dose: Receive NPH with each corticosteroid dose during the study duration (2-5 days).
  Low dose corticosteroids High dose corticosteroids Eating and 6a-8p 0.15 units NPH/kg 0.3 units NPH/kg NPO(nothing by mouth) or 8p-6a 0.1 units NPH/kg 0.2 units NPH/kg
  NPH: NPH given per study table based on steroid dose and patient weight in kg.
  Correction Factor: Given at 2 units per 50 mg/dl over 200 mg/dl and increased to 3 units/50 mg/dl over 200 if glucose rises to over 300 mg/dl. Administered qid during study duration.
- Total: Total of all reporting groups
Arm/Group | NPH With Corticosteroid Dose | Control | Total
Number analyzed (Participants) | 29 | 31 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 27 | 45
  >=65 years | 11 | 4 | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 17 | 32
  Male | 14 | 14 | 28
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 29 | 31 | 60

OUTCOME MEASURES:

1. Primary Outcome: Mean POC Glucose Level Between Groups
Description: Primary outcome measure was mean blood glucose levels measured pre-meal and at bedtime in study patients and controls for the duration of the intervention. Values shown are the overall mean point of care blood glucose.
Time Frame: Assessed from enrollment to discharge or enrollment to day five.
Measure: Mean (Standard Deviation); unit: mg/dl
Groups:
- NPH With Corticosteroid: Receive NPH with each corticosteroid dose during the study duration (2-5 days).
  Low dose corticosteroids High dose corticosteroids Eating and 6a-8p 0.15 units NPH/kg 0.3 units NPH/kg NPO(nothing by mouth) or 8p-6a 0.1 units NPH/kg 0.2 units NPH/kg
  NPH: NPH given per study table based on steroid dose and patient weight in kg.
  Correction Factor: Given at 2 units per 50 mg/dl over 200 mg/dl and increased to 3 units/50 mg/dl over 200 if glucose rises to over 300 mg/dl. Administered qid during study duration.
Arm/Group | NPH With Corticosteroid | Control
Number analyzed (Participants) | 29 | 31
mg/dl | 225 (87.2) | 266 (69.51)

2. Secondary Outcome: Episodes of Hypoglycemia Between NPH and Control Groups
Description: Hypoglycemia was defined as point of care glucose less than 70 mg/dL.
Time Frame: Glucose levels measured pre-meal, at bedtime, and during symptoms of hypoglycemia in study patients and controls for the duration of the intervention. Values shown represent cumulative episodes of hypoglycemia per group.
Measure: Number; unit: Hypoglycemic episodes.
Groups:
- NPH Insulin (Intervention Group): Receive NPH with each corticosteroid dose during the study duration (1-5 days).
  Low dose corticosteroids High dose corticosteroids Eating and 6a-8p 0.15 units NPH/kg 0.3 units NPH/kg NPO(nothing by mouth) or 8p-6a 0.1 units NPH/kg 0.2 units NPH/kg
  NPH: NPH given per study table based on steroid dose and patient weight in kg.
  Correction Factor: Given at 2 units per 50 mg/dl over 200 mg/dl and increased to 3 units/50 mg/dl over 200 if glucose rises to over 300 mg/dl. Administered qid during study duration.
- Control: Receive usual care with background insulin and correction factor for duration of study (1-5 days)
  Correction Factor: Given at 2 units per 50 mg/dl over 200 mg/dl and increased to 3 units/50 mg/dl over 200 if glucose rises to over 300 mg/dl. Administered qid during study duration.
Arm/Group | NPH Insulin (Intervention Group) | Control
Number analyzed (Participants) | 29 | 31
Hypoglycemic episodes. | 6 | 0

3. Other Pre Specified Outcome: Percentage of Point of Care Glucose Measurements Between 70 - 180 mg/dL
Description: Glucose levels measured pre-meal, at bedtime, and during symptoms of hypoglycemia in study patients and controls for the duration of the intervention. Values shown are the overall percentage of glucose measurements between 70 - 180 mg/dl.
Time Frame: From day 1 (day of enrollment) to day 5 (last day of study participation) or final day of hospitalization if less than 5 days. Point of care glucose was checked before breakfast, lunch, dinner, bed time and during symptoms of hypoglycemia.
Measure: Number; unit: Percentage of total measurements of gluc
Arm/Group | NPH Insulin (Intervention Group) | Control
Number analyzed (Participants) | 29 | 31
Percentage of total measurements of gluc | 33.1 | 19.2

4. Other Pre Specified Outcome: Incidence of Hyperglycemia Defined as Point of Care Glucose 180 - 300 mg/dL
Description: Glucose levels measured pre-meal, at bedtime, and during symptoms of hypoglycemia in study patients and controls for the duration of the intervention. Values shown are the overall percentage of glucose measurements 180 - 300 mg/dL.
Time Frame: as for outcome 3
Measure: Number; unit: Percentage of total measurements
Arm/Group | NPH Insulin (Intervention Group) | Control
Number analyzed (Participants) | 29 | 31
Percentage of total measurements | 42.1 | 45.3

5. Other Pre Specified Outcome: Incidence of Hyperglycemia Defined as Point of Care Glucose 300 - 400 mg/dl
Description: Glucose levels measured pre-meal, at bedtime, and during symptoms of hypoglycemia in study patients and controls for the duration of the intervention. Values shown are the overall percentage of glucose measurements 300 - 400 mg/dl.
Time Frame: as for outcome 3
Measure: Number; unit: Percentage of total measurements
Arm/Group | NPH Insulin (Intervention Group) | Control
Number analyzed (Participants) | 29 | 31
Percentage of total measurements | 16.9 | 27.0

6. Other Pre Specified Outcome: Incidence of Hyperglycemia Defined as Point of Care Glucose > 400 mg/dL
Description: Glucose levels measured pre-meal, at bedtime, and during symptoms of hypoglycemia in study patients and controls for the duration of the intervention. Values shown are the overall percentage of glucose measurements > 400 mg/dL.
Time Frame: as for outcome 3
Measure: Number; unit: Percentage of total measurements
Arm/Group | NPH Insulin (Intervention Group) | Control
Number analyzed (Participants) | 29 | 31
Percentage of total measurements | 5.9 | 8.5

7. Other Pre Specified Outcome: Difference in Length of Stay Between NPH and Control Group
Description: Time difference of hospitalization between the NPH and control groups.
Time Frame: Measured from the day of admission till the day of discharge
Population: Difference in mean length of stay between NPH group and usual care group
Measure: Mean (Full Range); unit: Days
Arm/Group | NPH Insulin (Intervention Group) | Control
Number analyzed (Participants) | 29 | 31
Days | 5.21 [1 to 5.25] | 5.23 [1 to 5.25]

8. Other Pre Specified Outcome: Mean Point of Care (POC) Glucose Level in Both Groups.
Description: The overall mean point of care glucose levels in the NPH group and control group on the first day of the study.
Time Frame: On day 1 of study enrollment. Point of care glucose was checked before breakfast, lunch, dinner, and bed time.
Population: Point of care glucose checked before breakfast, lunch, dinner, and bed time on day 1 of study enrollment. The numbers indicated below show the mean point of care (POC) glucose readings in the two groups on the first day of the study.
Measure: Mean (95% Confidence Interval); unit: mg/dL (mean values)
Arm/Group | NPH Insulin (Intervention Group) | Control
Number analyzed (Participants) | 29 | 31
mg/dL (mean values) | 246.9 [222.0 to 271.8] | 280.9 [257.6 to 304.1]

9. Other Pre Specified Outcome: Mean Point of Care (POC) Glucose Level in Both Groups.
Description: The overall mean point of care glucose levels in the NPH group and control group on the last day of the study.
Time Frame: On day 5 or last day of hospitalization (if less than 5 days) glucose level as measured by point of care glucose before breakfast, lunch, dinner and bed time.
Population: Point of care glucose checked before breakfast, lunch, dinner, and bed time on day 5 of study enrollment. The numbers indicated below show the mean point of care (POC) glucose readings in the two groups on the last day of the study.
Measure: Mean (95% Confidence Interval); unit: mg/dL (mean values)
Arm/Group | NPH Insulin (Intervention Group) | Control
Number analyzed (Participants) | 29 | 31
mg/dL (mean values) | 197.3 [170.9 to 223.6] | 253.5 [228.9 to 278.1]

10. Other Pre Specified Outcome: Correlation of C-peptide With Age
Time Frame: plasma C-peptide was measured once at the time of enrollment
Measure: Number; unit: correlation coefficient
Arm/Group | NPH Insulin (Intervention Group) | Control
Number analyzed (Participants) | 29 | 31
correlation coefficient | 0.197 | -0.226

11. Other Pre Specified Outcome: Correlation of C-peptide With BMI
Time Frame: Measured once at the time of enrollment
Measure: Number; unit: correlation coefficient
Arm/Group | NPH Insulin (Intervention Group) | Control
Number analyzed (Participants) | 29 | 31
correlation coefficient | 0.095 | 0.305

12. Other Pre Specified Outcome: Correlation of C-peptide With eGFR
Time Frame: Measured once at the time of enrollment
Measure: Number; unit: correlation coefficient
Arm/Group | NPH Insulin (Intervention Group) | Control
Number analyzed (Participants) | 29 | 31
correlation coefficient | -0.272 | -0.063

13. Other Pre Specified Outcome: Correlation of C-peptide With Serum Creatinine
Time Frame: Measured once at the time of enrollment
Measure: Number; unit: correlation coefficient
Arm/Group | NPH Insulin (Intervention Group) | Control
Number analyzed (Participants) | 29 | 31
correlation coefficient | 0.328 | -0.026

14. Other Pre Specified Outcome: Correlation of C-peptide With ALT
Time Frame: Measured once at the time of enrollment
Measure: Number; unit: correlation coefficient
Arm/Group | NPH Insulin (Intervention Group) | Control
Number analyzed (Participants) | 29 | 31
correlation coefficient | -0.358 | 0.436

15. Other Pre Specified Outcome: Correlation of C-peptide With Hemoglobin A1c
Time Frame: Measured once at the time of enrollment
Measure: Number; unit: correlation coefficient
Arm/Group | NPH Insulin (Intervention Group) | Control
Number analyzed (Participants) | 29 | 31
correlation coefficient | -0.325 | -0.251

16. Other Pre Specified Outcome: Correlation of C-peptide With Duration of Diabetes
Time Frame: Measured once at the time of enrollment
Measure: Number; unit: correlation coefficient
Arm/Group | NPH Insulin (Intervention Group) | Control
Number analyzed (Participants) | 29 | 31
correlation coefficient | -0.320 | -0.380

17. Other Pre Specified Outcome: Correlation of C-peptide With Plasma Glucose
Time Frame: Measured the time of enrollment
Measure: Number; unit: correlation coefficient
Arm/Group | NPH Insulin (Intervention Group) | Control
Number analyzed (Participants) | 29 | 31
correlation coefficient | 0.171 | -0.053

18. Other Pre Specified Outcome: Correlation of C-peptide With Length of Stay
Time Frame: Measured once at the time of enrollment
Measure: Number; unit: correlation coefficient
Arm/Group | NPH Insulin (Intervention Group) | Control
Number analyzed (Participants) | 29 | 31
correlation coefficient | -0.068 | -0.002

ADVERSE EVENTS:
Arm/Group | NPH With Corticosteroid | Control
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/31
Serious Adverse Events (participants affected / at risk) | 6/29 | 0/31
Other Adverse Events (participants affected / at risk) | 0/29 | 0/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NPH With Corticosteroid (N=29) | Control (N=31)
Hypoglycemia (Endocrine disorders) | 6 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No